CLINICAL TRIAL: NCT04292639
Title: Final Test Report for Vital USA Respiratory Rate Validation In Adults
Brief Title: Vital USA Respiratory Rate Validation In Adults
Acronym: RR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital USA, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR 2019-326
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Complication

STUDY DESIGN:
Intervention Model Description: The Vital Detect is a noninvasive device designed for spot-checking physiological parameters, such as Noninvasive Blood Pressure, Oxygen Saturation, Pulse Rate, Body Temperature, and Respiratory Rate. This device is a finger-cuff technology which is applicable for use at-home or in healthcare facilities in/on individuals 18 years of age and older. It may be used by the individual themselves or an operator. The Vital Detect is not intended for continuous monitoring or for use with high frequency surgical equipment. It is non transit-operable. The Vital USA Vital Detect is composed of a sensor head mounted on a base connected to a phone or computer via Vital Detect App which is free to download.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Respiratory Rate (Experimental): The purpose of this study is to conduct a Respiratory Rate accuracy validation comparing the Vital USA Vital Detect to an FDA cleared End Tidal Carbon Dioxide monitor Reference Standard (GE Datex-Ohmeda). This report documents exclusively the results of the Respiratory Rate accuracy performance for the Vital USA Vital Detect.
  Interventions: Device: The Vital Detect Pulse Oximeter

INTERVENTIONS:
Device: The Vital Detect Pulse Oximeter — The Vital Detect is a noninvasive device designed for spot-checking physiological parameters, such as Noninvasive Blood Pressure, Oxygen Saturation, Pulse Rate, Body Temperature, and Respiratory Rate. This device is a finger-cuff technology which is applicable for use at-home or in healthcare facilities in/on individuals 18 years of age and older. It may be used by the individual themselves or an operator. The Vital Detect is not intended for continuous monitoring or for use with high frequency surgical equipment. It is non transit-operable. The Vital USA Vital Detect is composed of a sensor head mounted on a base connected to a phone or computer via Vital Detect App which is free to download.
  Other Names: VitalDetect

SUMMARY:
Vital USA is dedicated to developing and applying innovative electronic medical solutions that improve patient care in multiple clinical settings. Vital USA is a manufacturer of a multi-parameter patient monitor that is intended to be used in a variety of medical settings including hospitals, medical offices and patients' homes.

DETAILED DESCRIPTION:
Purpose of Clinical Investigation Respiratory Rate is an important physiological measurement in the healthcare setting. End Tidal Carbon Dioxide (EtCO2) is considered to be the highest level of safety and accuracy in Respiratory Rate monitoring by the American Society of Anesthesiology and the American Association of Respiratory Care.

The purpose of this study was to conduct a Respiratory Rate accuracy validation comparing the Vital Detect to an FDA cleared End Tidal Carbon Dioxide monitor Reference Standard (GE Datex-Ohmeda).

Respiratory Rate is an important physiological measurement in the healthcare setting. End Tidal Carbon Dioxide (EtCO2) is considered to be the highest level of safety and accuracy in Respiratory Rate monitoring by the American Society of Anesthesiology and the American Association of Respiratory Care.

The purpose of this study was to conduct a Respiratory Rate accuracy validation comparing the Vital Detect to an FDA cleared End Tidal Carbon Dioxide monitor Reference Standard (GE Datex-Ohmeda).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is adult over 18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker
* Male or female of any race

Exclusion Criteria:

Subject is considered as being morbidly obese (defined as BMI >39.5)

* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
  * Cancer / chemotherapy
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark Laboratory Services, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The final study population consisted of 20 qualified healthy subjects, 10 males and 10 females, ranging in age from 18 to 52 yrs of any racial / ethnic background. Each subject understood the study and provided consent for participation by signing the Independent Review Board (IRB) approved Informed Consent Form prior to start of the test.
Pre-assignment Details: The subjects were healthy showing no evidence of significant medical problems as indicated by satisfactorily completing the health assessment form. Eligible subjects needed to meet all of the inclusion criteria and none of the exclusion criteria for participation.
Period: Overall Study
Arm/Group | Respiratory Rate
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 20 qualified healthy subjects, 10 males and 10 females, ranging in age from 18 to 52 years and of any racial / ethnic background. The subjects were healthy showing no evidence of significant medical problems as indicated by satisfactorily completing the health assessment form.
Groups:
- Respiratory Rate: This study was a comparative, single-center, non-randomized, parallel study, conducted on 20 subjects. The acceptance criteria in this study used a comparison of the Vital USA Vital Detect to a reference Respiratory Rate EtCO2 monitor. Testing was conducted under normal office environment conditions.
Arm/Group | Respiratory Rate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — All subjects between 18 to 52 years
  years | 29.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Equally counted 10 males and 10 females
  Participants
    Female | 10
    Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Any racial / ethnic background
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 19
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Fitzpatrick Scale [Count of Participants; unit: Participants]
  Type I Pale White Skin Blue/Green Eyes | 3
  Type II Fair Skin Blue Eyes | 12
  Type III Darker White Skin | 3
  Type IV Brown Skin | 0
  Type V Dark Brown Skin | 1
  Type VI Black Skin | 1
Weight [Mean (Standard Deviation); unit: Lbs] | 151.9 (25.9)
Height [Mean (Standard Deviation); unit: In] | 67.3 (3.9)
BMI [Mean (Standard Deviation); unit: lbs/sq.In.] | 23.5 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Rate Accuracy Validation for the Vital USA Vital Detect Monitor.
Description: The primary objective of this study was to compare the accuracy of device under test for the measurement of respiratory rate. The respiratory rate was measured simultaneously with EtCO2 (Reference) and the Vital USA Vital Detect monitor (Device Under Test).The endpoint of interest was accuracy as measured by the Accuracy root-mean-square (ARMS) difference between the Device Under Test (DUT) and the reference respiratory rate system (Ref) for all stable respiratory periods.
Time Frame: 20 Seconds
Population: The final study population consisted of 20 qualified healthy subjects, 10 males and 10 females, ranging in age from 18 to 52 years and of any racial / ethnic background.
Measure: Mean (Standard Deviation); unit: Breaths/Min
Groups:
- Respiratory Rate: The primary objective of this study was to compare the accuracy of device under test for the measurement of respiratory rate. The respiratory rate was measured simultaneously with EtCO2 (Reference) and the Vital USA Vital Detect monitor (Device Under Test).
Arm/Group | Respiratory Rate
Number analyzed (Participants) | 20
Breaths/Min | 1.39 (1.39)

ADVERSE EVENTS:
Time Frame: on the study date
Description: There were no serious adverse events or serious adverse device effects during the study.
Arm/Group | Respiratory Rate
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
There were no serious adverse events or serious adverse device effects during the study. There were no observed device deficiencies that could have led to serious adverse device effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT04292639/Prot_SAP_003.pdf